CLINICAL TRIAL: NCT03594981
Title: Adoptive Cord Blood ImmunotHerapy Using Expanded Cord Blood T Cells for EBV, CMV, BKV and Adenovirus Reactivation/Infection or ProphylaxiS
Brief Title: Adoptive Cord Blood Immunotherapy for EBV, CMV, BKV and Adenovirus Reactivation/Infection or Prophylaxis
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Catherine Bollard (Other)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor-Investigator, Catherine Bollard, Director, Center for Cancer and Immunology/ Center for Emerging Technologies in Immune Cell Therapies (CETI), Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHEERS
Record Dates: First submitted 2018-05-14; First posted 2018-07-23 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Viral Infection
MeSH Terms: conditions — Virus Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CMV/AdV /EBV/BKV specific T cells (Experimental): CMV/AdV /EBV/BKV specific T cells will be thawed and transferred to a syringe given by slow intravenous injection over 1-2 minutes. Three dose levels will be explored. The lowest dose level will be 1x107cells/m2 and the highest will be 5x107/m2.
  Interventions: Biological: CMV/AdV /EBV/BKV specific T cells

INTERVENTIONS:
Biological: CMV/AdV /EBV/BKV specific T cells — Each cohort of 2 patients will be treated and observed for 45 days for toxicity, dose escalation, and GvHD. The algorithm of sequentially adaptive EffTox trade-off-based design of Thall et al will be used to determine the dose for each cohort. If 1x107CTL/m2 results in unacceptable toxicity or efficacy, the study will be closed to accrual.

SUMMARY:
This Phase I-II dose-finding trial to determine the optimal dose of intravenous (IV) injection dose of donor-derived cytotoxic T lymphocytes (CTLs) specific for CMV, EBV, BKV and Adenovirus. A maximum of 36 patients will be treated in up to 18 cohorts each of size 2, with the first cohort treated at the lowest dose level 1, all successive doses chosen by the EffTox method, and no untried dose level skipped when escalating.

The scientific goal of the trial is to determine an optimal IV-CTL cell dose level among the three doses 1.0x107cells/m2, 2 x107cells/m2 and 5x107cells/m2., hereafter dose levels 1, 2, 3. Dose-finding will be done using the sequentially adaptive EffTox trade-off-based design of Thall et al.

DETAILED DESCRIPTION:
This Phase I-II dose-finding trial to determine the optimal dose of intravenous (IV) injection dose of donor-derived cytotoxic T lymphocytes (CTLs) specific for CMV, EBV, BKV and Adenovirus. A maximum of 36 patients will be treated in up to 18 cohorts each of size 2, with the first cohort treated at the lowest dose level 1, all successive doses chosen by the EffTox method, and no untried dose level skipped when escalating.

The scientific goal of the trial is to determine an optimal IV-CTL cell dose level among the three doses 1.0x107cells/m2, 2 x107cells/m2 and 5x107cells/m2., hereafter dose levels 1, 2, 3. Dose-finding will be done using the sequentially adaptive EffTox trade-off-based design of Thall et al. To implement the design's model using the latest EffTox version 4.0.12 program, doses will coded numerically to be 1, 2, 3.

CMV/AdV /EBV/BKV specific T cells will be thawed and given or thawed and diluted into a total volume of 10 mL of Plasmalyte A by slow intravenous injection over 1-2 minutes. This is a traditional Phase I dose escalation study of a single infusion of CMV/AdV/EBV/BKV-specific CTLs to patients at risk for CMV and EBV reactivation and Adenoviral and BK virus infection after umbilical cord blood transplantation. Three dose levels will be explored. The lowest dose level will be 1x107cells/m2 and the highest will be 5x107/m2. There will be 2-6 patients at each dose level (depending on toxicity) following the scheme below. The decision on whether it is safe to escalate to next dose level or not will be made after at least two patients in each dose level have finished their 45-days toxicity follow up. If the first two patients have not finished their 45 days follow-up, up to 2 additional incoming patients can be enrolled at the current dose level. In addition, we will give the option of administering 2 additional doses (at the same dose level), 28 days after the first infusion of the same dose, in subjects who have a partial response after one dose or who have received other therapy that may affect the persistence or function of the infused CTL in vivo. If there are no toxicities and immunological efficacy is not seen at any dose, then the doses will be further escalated after additional local and federal approval.

Dose Levels and Dosing Schedule

Dose Level CTL Dose Given from Day +30 post SCT

1. 1x107/m2
2. 2.0x107/m2
3. 5x107/m2

Escalation of Multi-virus-specific CTL infusions

CMV/AdV/EBV/BKV CTL will be given from day +30 either as prophylaxis or treatment for CMV, EBV, BK and/or adenovirus infection. If the patient has viral reactivation or evidence of CMV/EBV/AdV/BKV disease (e.g. pneumonitis, gastroenteritis and/or retinitis or Post Transplant Lymphoproliferative Disorder (PTLD) or hemorrhagic cystitis the CTL can be given with concurrent antiviral pharmacotherapy.

A dose escalation scheme utilizing cohorts of two patients will be used

Each cohort of 2 patients will be treated and observed for 45 days for toxicity, dose escalation, and GvHD. The algorithm described in Section 9 will be used to determine the dose for each cohort. If 1x107CTL/m2 results in unacceptable toxicity or efficacy, the study will be closed to accrual.

The Optimal Dose of Infused CMV/AdV/EBV/BKV-Specific CTL

After all patients in the trial have been evaluated, the optimal dose of infused CMV/AdV/EBV-specific CTL will be determined by the algorithm using the sequentially adaptive EffTox trade-off-based design of Thall et al.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria at the Time of Procurement

* Pediatric and adult patients (there are no lower and upper age limits for patients) with malignant or nonmalignant diseases who are candidates for transplant.
* Patients must have a CB unit (or units) matched with the patient at 4, 5, or 6/6 HLA class I (serological) and II (molecular) antigens. The unit selected for CTL expansion must be either:

  1. be cryopreserved in two fractions, with a minimum of 2.5x107 total nucleated cells (TNC) per kg pre-thaw in the fraction which will be used for the primary transplant. The remaining fraction will be used to generate the CTLs to give at day 30 or beyond as described below. OR
  2. be cryopreserved with a cell dose that totals > 3x10e7 TNC per kg pre thaw. On thaw, 20% of the total volume will be used for CTL manufacture to give at day 30 or beyond and the remaining 80% will be used for the primary transplant.
  3. For recipients of double CBT, if possible both CB units should be cryopreserved in two fractions and T-cells will be made from both units if possible.

Inclusion Criteria at the Time of CTL Infusion

* Recipients of at least one unmanipulated cord blood unit as described above (i.e. from a HLA matched or mismatched unrelated donor) transplant at risk for or with CMV/Adenoviral/BKV and/or EBV infection or reactivation.
* Lansky/Karnofsky scores ≥60
* Absolute neutrophil count (ANC) greater than 500/u
* No evidence of GVHD > Grade II at time of enrollment
* Life expectancy > 30 days
* Absence of severe renal disease (Creatinine < 3x normal for age)
* Absence of severe hepatic disease. Direct bilirubin must be < 3 mg/dl and AST < 5x upper limit of normal
* Patient must be at least 30 days post transplant to be eligible to receive CTL
* Written informed consent and/or signed assent line from patient, parent or guardian

Exclusion Criteria:

Exclusion Criteria at the Time of Procurement

* Pregnant or lactating
* Patients with active central nervous system disease
* Patients with Karnofsky performance status <70%
* Patients with grade 3 or 4 or primary myelofibrosis
* Patients with suitable related donors Exclusion Criteria at the Time of CTL Infusion
* Pregnant or lactating
* Patient on Fi02 of >60%
* Unable to wean steroids to ≤0.5 mg/kg/day prednisone or equivalent
* Patients with Grade 3 hyperbilirubinemia
* Patients with other uncontrolled infections (except CMV and/or adenovirus and/or EBVemia and/or BK viruria/viremia). For bacterial infections, patients must be receiving definitive therapy and have no signs of progressing infection for 72 hours prior to enrollment. For fungal infections patients must be receiving definitive systemic anti-fungal therapy and have no signs of progressing infection for 1 week prior to enrollment. Progressing infection is defined as hemodynamic instability attributable to sepsis or new symptoms, worsening physical signs or radiographic findings attributable to infection. Persisting fever without other signs or symptoms will not be interpreted as progressing infection.
* Patients with less than 50% donor chimerism in either peripheral blood or bone marrow or patients with relapse of original disease
* Patients who have received investigational (IND) product within 28 days of screening for CTL infusion under this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2018-01-24 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants with investigational product-related adverse events as assessed by CTCAE v4.03 | 45 days for toxicity
  The study will determine the optimal dose of intravenous injection of donor-derived cytotoxic T lymphocytes (CTLs) specific for CMV, EBV, Adenovirus and BK virus( BKV) given to patients with or at risk for CMV, EBV, BK virus and adenovirus infection after cord blood transplant. The safety will be assessed by investigational product-related adverse events as per CTCAE v4.03.

SECONDARY OUTCOMES:
Impact of CMV/AdV /EBV/BKV specific T cells will be measured by existence of cells in the system. | 12 months
  To evaluate the impact of CTLs on CMV/AdV /EBV/BKV -specific T-lymphocyte immune reconstitution. The impact will be evaluated by the number of months/years of cell survival.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Children's National Health System, Washington D.C., District of Columbia
  - M.D. Anderson Cancer Center (MDACC), Houston, Texas

IPD SHARING:
Plan to Share IPD: No